CLINICAL TRIAL: NCT05449600
Title: Thermotape High-adhesion Medical Tape Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Washington Institute for Translational Health Science (UL1 TR002319) (Unknown)
Responsible Party: Principal Investigator, Eric Seibel, Research Professor: Mechanical Engineering, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: STUDY00014704; U01HL152401 (NIH)
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Skin Injury

STUDY DESIGN:
Intervention Model Description: Tegaderm™ tape, Kind™ tape, and Thermotape will be applied to both forearms for 24 hours. Afterwards, one forearm will have the tapes removed normally, without any intervention. The other forearm will have the tapes removed after heat is applied, using a heatpack.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participant (Experimental): Tegaderm™ tape, Kind™ removal tape, and Thermotape will be applied to both of the participant's forearms.
  Interventions: Device: Thermotape; Device: Tegaderm; Device: Kind
- Researcher (No Intervention)

INTERVENTIONS:
Device: Thermotape — Thermotape will be applied along the left and right forearm. One piece of tape, one inch wide by two inches long, will be applied to each arm. The location the tape, when applied, will be randomized. Altogether, two pieces of this particular tape will be applied, one to each forearm.
  Arms: Participant
Device: Tegaderm — Tegaderm™will be applied along the left and right forearm. One piece of tape, one inch wide by two inches long, will be applied to each arm. The location the tape, when applied, will be randomized. Altogether, two pieces of this particular tape will be applied, one to each forearm.
  Arms: Participant
Device: Kind — Thermotape will be applied along the left and right forearm. One piece of tape, one inch wide by two inches long, will be applied to each arm. The location the tape, when applied, will be randomized. Altogether, two pieces of this particular tape will be applied, one to each forearm.
  Arms: Participant

SUMMARY:
This objective of this study is to compare the safety and performance of Thermotape compared to Tegaderm™ tape and Kind™ tape over the course of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be between 18 to 25 years of age.

Exclusion Criteria:

* Participants with history of eczema or medical related skin injuries (MARSI), allergic to adhesives, and/or have a wound or rash on their skin will be excluded.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Pain Experienced by Tape Removal | Each removal and assessment would take at maximum 5 minutes.
  A 0 to 10 point Wong-Baker FACES Pain Rating Scale will be used to quantify the pain felt by the subject when each tape is removed. A score of 0 represents no pain experienced by removal, while 10 represents severe pain experienced during tape removal.
Skin Irritation | Subjects will wait approximately 15 minutes before leaving, to ensure that irritation has occurred.
  Redness of the skin will be examined after tape is removed.

SECONDARY OUTCOMES:
Skin cells | The removal of each tape will take a maximum of 2 minutes.
  The skin cells removed from the skin during tape removal will be quantified. This will be performed by staining the tape and counting the cells under a light microscope.
Wear | The removal of each tape will take a maximum of 2 minutes.
  The condition of the tape after 24 hours will be examined. A 0 to 7 point scale will be used to quantify the wear, with 0 representing the maximum amount of wear, where the tape strip is no longer attached, while 7 represents little to no wear, with all corners of the tape fully adhered.
Hair Follicles | The removal of each tape will take a maximum of 2 minutes.
  Arm hair removed from tape removal will be quantified.
Trans-epidermal Water Loss | The removal of each tape will take a maximum of 2 minutes.
  Water loss experienced by the epidermis after tape removal will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Seibel, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

DOCUMENTS (3):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT05449600/Prot_003.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT05449600/SAP_001.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT05449600/ICF_002.pdf